CLINICAL TRIAL: NCT01422824
Title: An Observational. Non-interventional Study to Observe the Safety and Efficacy of MIRCERA in the Treatment of Chronic Renal Anemia in Maintenance ESA Treated Patients on Haemodialysis (STABILE)
Brief Title: An Observational Study of Mircera (Methoxy Polyethylene Glycol-Epoetin Beta) as Maintenance Treatment in Patients With Chronic Renal Anemia on Haemodialysis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25067
Record Dates: First submitted 2011-08-23; First posted 2011-08-24 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-02

CONDITIONS: Anemia, Kidney Disease, Chronic
MeSH Terms: conditions — Anemia; Kidney Diseases; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This prospective observational study will evaluate the safety and efficacy of Mircera (methoxy polyethylene glycol-epoetin beta) in patients with chronic renal anemia on haemodialysis in maintenance ESA treatment. Data will be collected from patients receiving once monthly Mircera according to standard of care and local labelling during 12 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Stage IV chronic kidney disease, on haemodialysis
* Chronic renal anemia, on maintenance ESA treatment
* Hemoglobin concentration between 10.0 an 12 g/dL
* Continuous maintenance epoetin therapy with the same dosing interval during the previous month

Exclusion Criteria:

* Contraindications to ESA treatment (e.g. hypersensitivity, non-controlled hypertension)
* Hemoglobinopathies (e.g. homozygous sickle-cell disease, thalassemia of all types)
* Anemia due to hemolysis, pure red cell aplasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic renal anemia on haemodialysis in maintenance ESA treatment
Sampling Method: Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2010-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- North Macedonia (6):
  - Delcevo
  - Prilep
  - Shtip
  - Skopje
  - Struga
  - Strumica

RESULTS

PARTICIPANT FLOW:
Groups:
- Mircera: Participants received Mircera® (methoxy polyethylene glycol-epoetin beta) according to the standard practice in line with current summaries of product characteristics (SPCs)/local labeling.
Period: Overall Study
Arm/Group | Mircera
Started | 185
Treated | 184
Completed | 147
Not Completed | 38
Not completed — Case record form not evaluated | 1
Not completed — Lost to Follow-up | 37

BASELINE CHARACTERISTICS:
Population: Safety population included all treated participants.
Groups:
- Mircera: Participants received Mircera® (methoxy polyethylene glycol-epoetin beta) according to the standard practice in line with current SPCs/local labeling.
Arm/Group | Mircera
Number analyzed (Participants) | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 106

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: AE: any unfavorable and unintended sign, symptom, or disease associated with use of study drug, regardless of relation to study drug. Pre-existing conditions that worsened and laboratory or clinical tests that resulted in change in treatment or discontinuation from study drug were reported as AEs. Serious AE (SAE): resulted in death, life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was congenital anomaly/birth defect, or was medically significant. Any AE included participants with both serious and non-serious AEs.
Time Frame: Up to 12 months
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Mircera
Number analyzed (Participants) | 184
participants
  Any AE | 49
  SAE | 22

2. Secondary Outcome: Hemoglobin Levels
Time Frame: Baseline; Weeks 8, 16, 24, 48
Population: Efficacy intent-to-treat population included all treated participants. Here, 'n' signifies the number of participants with available data for hemoglobin at specified visits.
Measure: Mean (Standard Deviation); unit: gram per liter
Arm/Group | Mircera
Number analyzed (Participants) | 184
gram per liter
  Baseline (n=184) | 110.3 (8.671274)
  Week 8 (n=179) | 110.8 (13.31517)
  Week 16 (n=155) | 111.3 (14.97250)
  Week 24 (n=161) | 111.2 (14.93382)
  Week 48 (n=130) | 111.2 (13.5594)

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: Safety population.
Arm/Group | Mircera
Serious Adverse Events (participants affected / at risk) | 22/184
Other Adverse Events (participants affected / at risk) | 14/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera (N=184)
Decreased hemoglobin (Blood and lymphatic system disorders) | 1
Myocardial infarction (Cardiac disorders) | 4
Chest pain - cardiac (Cardiac disorders) | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Death (General disorders) | 5
Cholecystitis (Hepatobiliary disorders) | 1
Vascular access thrombosis (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis with melena (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic event (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera (N=184)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.